CLINICAL TRIAL: NCT01662414
Title: Effect of Undenatured Cysteine-Rich Whey Protein Isolate (HMS 90®) in Patients With Parkinson's Disease: Changes in Biomarkers of Oxidative Stress, Profiles of Plasma Amino Acids and Their Derivatives and Brain Function
Brief Title: Effect of Undenatured Cysteine-Rich Whey Protein Isolate (HMS 90®) in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 53653
Record Dates: First submitted 2012-08-07; First posted 2012-08-10 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Parkinson Disease; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Neurodegenerative Diseases | interventions — Whey Proteins; Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- HMS 90® (Active Comparator)
  Interventions: Dietary Supplement: Whey protein
- Placebo (Soy protein) (Placebo Comparator)
  Interventions: Dietary Supplement: Soy protein

INTERVENTIONS:
Dietary Supplement: Whey protein — 1 sachect (10 g) 2times/ day
  Arms: HMS 90®
Dietary Supplement: Soy protein — 1 sachect (10g) 2times/day
  Arms: Placebo (Soy protein)

SUMMARY:
This is a double-blind, placebo-controlled, Phase IV trial , comparing HMS 90® versus placebo (soy protein) as add-on (adjuvant) therapy in subjects with idiopathic Parkinson's Disease.

The principal objective is to evaluate the changes in biomarkers of oxidative stress and,plasma amino acids, as well as improvement of clinical symptoms and brain function

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with Idiopathic Parkinson's Disease
2. Subjects who are willing and able to participate in the trial and has provided written, informed consent.

Exclusion Criteria:

1. Subjects who are allergic to Whey protein (HMS 90®).
2. Subjects who are treated with chemotherapy .
3. Subjects with any history of neurodegenerative diseases, e.g., Alzheimer's disease.
4. Subjects with history of diabetes. 4.5. Subjects with abnormal liver function test

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Biomarkers of oxidative stress, i.e., plasma glutathione (reduced and oxidized forms), urinary 8-hydroxydeoxyguanosine, and urinary total antioxidant status | 6 months
Concentrationsrofiles of plasma amino acids and their derivatives Brain function by PET-Scan | 6 months

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) Section III (motor) score change from baseline to week 24 | 6 months
Unified Parkinson's Disease Rating Scale (UPDRS) Section II (ADL) score change baseline to week 24 | 6 months
• Clinical Global impression (CGI) - Change scale score, change from baseline to week 24 | 6 months
• Clinical Global impression (CGI) - Severity scale score change from baseline to week 24 | 6 months
• Parkinson's Disease quality of life questionnaire score change from baseline to week 24 | 6 months
Nutrition Questionnaire score change baseline to week 24 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Roongroj Bhidayasiri, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University Hospital, Pathumwan, Bangkok, Thailand